CLINICAL TRIAL: NCT03220464
Title: Early Diagnosis of Active Tuberculosis Using Ultra Low-dose Chest CT to Predict Progression to Active Tuberculosis Among Contacts
Brief Title: Early Diagnosis of Active Tuberculosis Using Ultra Low-dose Chest CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1704-157-849
Record Dates: First submitted 2017-06-25; First posted 2017-07-18 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Tuberculosis, Pulmonary; Latent Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Latent Tuberculosis | interventions — X-Rays; Interferon-gamma Release Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Close contacts of active pulmonary tuberculosis patients (Experimental): One arm study of conducting ULDCT, chest x-ray, and IGRA
  Interventions: Radiation: Ultra low dose chest computed tomography (ULDCT); Radiation: Chest X-ray; Diagnostic Test: Interferon-gamma Release Assay (IGRA)

INTERVENTIONS:
Radiation: Ultra low dose chest computed tomography (ULDCT) — Participants in the study will receive ULDCT at enrollment, after 3-month visit, and after 12-month visit.
Radiation: Chest X-ray — Participants in the study will receive chest x-ray at enrollment, after 3-month visit, and after 12-month visit.
  Other Names: Chest radiograph
Diagnostic Test: Interferon-gamma Release Assay (IGRA) — Participants in the study will receive IGRA test at enrollment, after 3-month visit, and after 12-month visit. About 11mL of blood will be drawn from the participants for test of T-SPOT®.TB test and QuantiFERON test.

SUMMARY:
The aim of this study is to evaluate ultra low dose chest computed tomography (ULDCT) for early diagnosis of active tuberculosis in cohort of close contacts of active pulmonary tuberculosis for 1 year follow up

DETAILED DESCRIPTION:
The early diagnosis of active tuberculosis in close contacts have not yet been established. To evaluate the early detection of active pulmonary tuberculosis using ULDCT, the investigators will establish the observational cohort of close contacts living in the same space with active pulmonary tuberculosis. Participants will visit our center at enrollment, after 3 months, and 12 months and will be received ULDCT, chest X-ray and Interferon-gamma assays at each visit. One chest radiologist will interpret findings of ULDCT and chest X-ray.

Patients diagnosed with active tuberculosis will be excluded from the study and treated based on World Health Organization guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Close contacts of active pulmonary tuberculosis
* Family members of active TB patient who has lived together for more than one month, or work colleagues of active TB patient who has been working in the same office for more than 8 months
* Participants who received explanation of the research plan, understands and writes agreement.

Exclusion Criteria:

* Vulnerable subjects with mental retardation or severe mental illness
* Patients who could not receive chest CT
* Pregnancy
* Close contacts who diagnosed active pulmonary tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of active pulmonary tuberculosis | For a year
  Active pulmonary tuberculosis defined by WHO guidelines for treatment of drug-susceptible tuberculosis and patient care (2017 update)

SECONDARY OUTCOMES:
Prevalence of active pulmonary tuberculosis at enrollment | Baseline
  Active pulmonary tuberculosis defined by WHO guidelines for treatment of drug-susceptible tuberculosis and patient care (2017 update)
Prevalence of latent tuberculosis at enrollment | Baseline
  Latent tuberculosis defined by guidelines on the management of latent tuberculosis infection
Change of ultra low dose chest CT findings in latent tuberculosis patients | Baseline, 3-month follow-up, and 12-month follow-up
  Serial comparison analysis of CT findings in latent tuberculosis patients who diagnosed latent tuberculosis based on IFN-gamma assay

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization, and Stop TB Initiative (World Health Organization). Treatment of tuberculosis: guidelines. World Health Organization, 2010.
- [Background] Guidelines on the Management of Latent Tuberculosis Infection. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK293818/ PMID 25973515
- [Result] Lee SW, Jang YS, Park CM, Kang HY, Koh WJ, Yim JJ, Jeon K. The role of chest CT scanning in TB outbreak investigation. Chest. 2010 May;137(5):1057-64. doi: 10.1378/chest.09-1513. Epub 2009 Oct 31. PMID 19880906
- [Result] Piccazzo R, Paparo F, Garlaschi G. Diagnostic accuracy of chest radiography for the diagnosis of tuberculosis (TB) and its role in the detection of latent TB infection: a systematic review. J Rheumatol Suppl. 2014 May;91:32-40. doi: 10.3899/jrheum.140100. PMID 24788998
- [Result] Lew WJ, Jung YJ, Song JW, Jang YM, Kim HJ, Oh YM, Lee SD, Kim WS, Kim DS, Kim WD, Shim TS. Combined use of QuantiFERON-TB Gold assay and chest computed tomography in a tuberculosis outbreak. Int J Tuberc Lung Dis. 2009 May;13(5):633-9. PMID 19383198
- [Result] Fujikawa A, Fujii T, Mimura S, Takahashi R, Sakai M, Suzuki S, Kyoto Y, Uwabe Y, Maeda S, Mori T. Tuberculosis contact investigation using interferon-gamma release assay with chest x-ray and computed tomography. PLoS One. 2014 Jan 14;9(1):e85612. doi: 10.1371/journal.pone.0085612. eCollection 2014. PMID 24454900
- [Result] Sloot R, Schim van der Loeff MF, Kouw PM, Borgdorff MW. Risk of tuberculosis after recent exposure. A 10-year follow-up study of contacts in Amsterdam. Am J Respir Crit Care Med. 2014 Nov 1;190(9):1044-52. doi: 10.1164/rccm.201406-1159OC. PMID 25265362
- [Result] Fox GJ, Barry SE, Britton WJ, Marks GB. Contact investigation for tuberculosis: a systematic review and meta-analysis. Eur Respir J. 2013 Jan;41(1):140-56. doi: 10.1183/09031936.00070812. Epub 2012 Aug 30. PMID 22936710